CLINICAL TRIAL: NCT07164885
Title: Phase II/III Randomized Clinical Trial of Radiosensitivity-Assisted Personalized Adaptive RadioTherapy (RAPART) in Locally Advanced Non-small Cell Lung Cancer Patients
Brief Title: RAPART in Locally Advanced Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jin jianyue, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCOG0058
Record Dates: First submitted 2025-06-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): RAPART technology
  Interventions: Radiation: Radiosensitivity-Assisted Personalized Adaptive Radiotherapy Technology（RAPART)）
- conventional radiotherapy (Active Comparator): conventional radiotherapy 2Gy/F
  Interventions: Radiation: Conventional radiotherapy

INTERVENTIONS:
Radiation: Radiosensitivity-Assisted Personalized Adaptive Radiotherapy Technology（RAPART)） — RAPART technology is a special combination of ART and RAPRT, with a total course limit of no more than 30 exposures. The entire course of treatment can be divided into two stages: the first stage is completely the same as the conventional radiotherapy group, with a total of 23 doses of 2 Gy per session. The second stage is the combination of ART and PAPRT. ART uses a CT or PET/CT localization simulation to be performed again during the course of treatment (usually after completing the first part of 17-19 exposures) to generate a new adaptive plan, and after completing the first stage of 23 exposures, treatment is carried out according to the new adaptive plan. RAPAT uses ERCC1/2 biomarkers to predict the patient's radiation sensitivity and determine individualized radiation dose accordingly. ERCC1/2 biomarkers divided patients into 5 different radiosensitivity groups, corresponding to 5 different radiation doses (74, 66, 62, 54, and 50 Gy).
  Arms: Experiment
Radiation: Conventional radiotherapy — conventional radiotherapy
  Arms: conventional radiotherapy

SUMMARY:
This is a Phase II/III randomized clinical trial of Radiosensitivity-Assisted Personalized Adaptive Radiotherapy Technology (RAPART) in locally advanced non-small cell lung cancer patients. The main objective is to test the overall improvement of overall survival (OS), progression free survival (PFS), and local progression free survival (LPFS) of unresectable stage III NSCLC under standard and non-standard mixed treatment conditions compared to conventional 60Gy radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult research participants, aged over 18 years old;
* Non small cell lung cancer that requires pathological confirmation;
* All stage 3 unresectable non-small cell lung cancer, including stage correction after MDT and stage downgrading after treatment (4 → 3), and stage upregulation due to disease progression (2 → 3);
* ECOG physical condition is 0-2;
* In addition to study participants who have not received any treatment, study participants who have undergone surgery, chemotherapy, immunotherapy, and targeted therapy are also eligible for enrollment.

Exclusion Criteria:

* Prisoners who are not convenient for close clinical follow-up;
* Study participants with contraindications to radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 911 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
progression-free survival | From enrollment to 3 years after the end of treatment
Toxic events | From enrollment to 3 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No